CLINICAL TRIAL: NCT00772863
Title: The Evaluation of Efficacy and Safety of Subsequent Cisplatin and Docetaxel Regimen In The First Line Treatment of Advanced Epithelial Ovarian Cancer
Brief Title: Efficacy and Safety of Subsequent Cisplatin and Docetaxel in Ovarian Cancer
Acronym: Tax-Over
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976I_6012
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel and cisplatin — 4 cycles Cisplatin 100 mg/m2 at every 3 weeks, after Cisplatin 4 cycles of docetaxel 100mg/m2 at every 3 weeks

SUMMARY:
The purpose of this study is to assess the efficacy and the safety of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed, optimally debulked stage III-IV epithelial ovarian cancer excluding clear cell histology.
* ECOG Performance Status is 0-2
* No prior chemotherapy for this malignancy,
* Acceptable hematological profile (as defined by a leukocyte count ≥ 3000/mm3, a platelet count ≥ 100.000mm3 and Hb ≥ 9g/100mL), and adequate renal function (as defined by serum creatinine ≤ 1.5mg/dl or creatinine clearance by formulation ≥ 60 mL/min), and hepatic function (as defined by bilirubin ≤ 1.5 x maximum normal value even with hepatic metastasis; transaminases (ALT, AST) ≤ 1.5 x maximum normal value; alkaline phosphatase ≤ 2.5 x maximum normal value, except in case of a bone metastasis)

Exclusion Criteria:

* Concomitant use of another anti-cancer therapy
* Unstable medical condition that makes the patient unable to take part in a clinical study (congestive heart failure, serious arrythmia, uncontrolled diabetes mellitus), history of myocardial infarction within last 3 months, massive pleural, peritoneal or pericardial effusion; or presence of serious uncontrolled infection.
* Presence of other tumours different from basal cell carcinoma of the skin.
* Pregnancy or breastfeeding. In women of childbearing potential and in men, an adequate contraceptive method must be used
* Social or psychological condition that render the patient inadequate for the follow-up of the study
* Contraindication for any of the study drugs (e.g. history of hypersensitivity to any of the ingredients of the study drugs)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2003-09; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Efficacy by response rate according to RECIST criteria and safety | After the 2nd cycle, 4th cycle and 8th cycle and at the follow up period

SECONDARY OUTCOMES:
Time to disease progression or relapse | Until progression througout the study
Survival time | Througout the study
Quality of life based on the questionnaire EORTC QLQ-C30 filled by the patients | Prior to entry, after completion of treatment and at the first follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, MD, Study Director — Sanofi
Locations (1):
- Sanofi aventis administrative office, Istanbul, Turkey (Türkiye)